CLINICAL TRIAL: NCT02186938
Title: Does the Intraoperative Use of the FloTrac Device to Guide Fluid and Vasopressor Management Affect Postoperative Morbidity in Patients Receiving a Head and Neck Microvascular Free Tissue Transfer
Brief Title: A Prospective Study Evaluating the Use of Intraoperative Stroke Volume Variation Via the FloTrac Device to Guide Fluid and Vasopressor Management in Head and Neck Free Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ENT FloTrac
Record Dates: First submitted 2014-06-20; First posted 2014-07-10 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer; Patients Requiring a Free Flap Surgery
Keywords: head and neck cancer; patients requiring a free flap surgery
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Arterial line (radial, femoral, dorsalis pedis, or brachial), central line for access when needed, intubation vs tracheostomy, general anesthesia. We currently use stroke-volume variability monitoring (FloTrac) in all patients using the arterial line placed for blood pressure monitoring.
- Treatment (Experimental): The study will use a treatment algorithm for patients in the treatment group. This algorithm will aim to maintain a near-normal blood pressure and use goal directed therapy to achieve this. Currently the standard of care is to use IV fluid exclusively in these patients and anesthesia providers everywhere have been challenging that treatment plan. Our algorithm has an iterative approach assessing volume status, cardiac output and vascular tone in order, with interventions specified for each. Individual treatments have been proven safe and effective in this population, we believe this sequence may be the best current management system. By avoiding excessive fluid administration we expect to decrease ICU length of stay due to the comorbidities caused (pulmonary edema, bowl edema, glycocalyx damage).
  Interventions: Device: FloTrac

INTERVENTIONS:
Device: FloTrac
  Arms: Treatment

SUMMARY:
This study aims to investigate whether the intraoperative use of the FloTrac device to guide fluid and vasopressor management during head and neck free flap surgery improves postoperative outcome. Primary postoperative outcome is length of hospital stay. Secondary postoperative outcomes include days in ICU, days on ventilator, presence of postoperative pulmonary edema, need for postoperative vasopressors or transfusions, 30 day flap complication rate, inpatient postoperative cardiorespiratory complications/events, and overall 30 day flap failure rate.

DETAILED DESCRIPTION:
Few animal models have shown that intravenous vasopressor administration (including use of pure alpha agonists such as phenylephrine) can decrease blood flow to free musculocutaneous flaps (1-3). This has led to a dogmatic belief that all vasopressors should be avoided intraoperatively during a microvascular free flap reconstruction regardless of patient hemodynamics, even though there is little published evidence that pressors negatively affect free flap outcome (4). As a result, these patients often receive generous amounts of fluids during their intraoperative course to combat periods of hypotension. However, patients receiving head and neck free tissue transfers tend to be older with serious comorbidities related to long term tobacco use such as significant cardiovascular and pulmonary disease. Thus, they often exhibit intraoperative hemodynamic lability with periods of hypotension that may not necessarily be related to hypovolemia. Consistently treating periods of hypotension with more intravenous fluids can lead to serious postoperative complications such as graft failure (4), pulmonary edema, and congestive heart failure. In fact, we have just completed a retrospective review of 248 patients over a 34 month period that received a head and neck free tissue transfer; we discovered that a 1ml/kg/hr increase in intraoperative fluid administration significantly increased 30 day flap complication rate while intraoperative administration of vasopressors did not affect 30 day flap complication or 30 day failure rate.

The FloTrac device is an approved and validated medical device that analyzes the arterial pressure waveform to calculate a stroke volume variation. This stroke volume variation can be used to better guide intraoperative patient therapy with regard to need for fluid vs. pressor management during periods of intraoperative hypotension (5). The use of the FloTrac device for goal directed therapy has been investigated in major abdominal surgery and found to decrease length of hospital stay and complication rate in this surgical population (5-6). Thus, it is possible that the intraoperative use of the FloTrac device can better guide anesthesia providers to provide the necessary therapy for intraoperative hypotension in patients undergoing head and neck freet tissue transfer, thus improving postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* adults requiring "free flap" tissue reassignment surgery for head and neck cancer at either MUSC or Vanderbilt Medical Center

Exclusion Criteria:

* Patients < 55kg or > 140 kg based on literature regarding accuracy of flotrac.
* Patients with sustained intraoperative dysrrhythmias based on literature regarding accuracy of flotrac (ie, atrial flutter, atrial fibrillation).
* Patients with diagnosed NYHA class III-IV failure or documented EF < 30%
* Patients with pulmonary disease preventing administration of goal tidal volumes without excessive inspiratory pressures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Reeves, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: FloTrac device was used to manage blood pressure during surgery.
- Control Group: FlotTrac device was not used. Blood pressure of the control group was managed with standard methods.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 47 (2012) | 47
Completed | 38 | 44
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [22 to 81] | 57.6 [18 to 84] | 57.7 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: ICU Stay
Description: The primary outcome is length of ICU stay.
Time Frame: Participants were assessed from entry into ICU until departure.
Measure: Mean (Full Range); unit: hours
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 47 | 47
hours | 33.7 [12.5 to 102] | 58.3 [2 to 207]

2. Secondary Outcome: Number of Participants Requiring a Ventilator
Description: The secondary outcome is decreasing patient morbidity by comparing the number of patients on the ventilator
Time Frame: The number of participants requiring a ventilator after surgery.
Measure: Number; unit: participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 47 | 47
participants | 9 | 18

ADVERSE EVENTS:
Time Frame: Participants were followed for one year following their surgery.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes